CLINICAL TRIAL: NCT03015415
Title: A Prospective Randomized Controlled Trial of Open Arthrolysis Versus Non-surgical Treatment for Elbow Stiffness
Brief Title: The Posttraumatic Elbow Stiffness Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, César Luiz Betoni Guglielmetti, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Clbguglielmetti
Record Dates: First submitted 2017-01-05; First posted 2017-01-10 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Elbow Joint Contracture; Elbow Flexion Contractures; Elbow Injury; Elbow Osteoarthritis
Keywords: elbow; posttraumatic stiffness; elbow contractures; stiff elbow; dynamic orthoses; Dynamic splint; Rehabilitation; Splint; Effectiveness of bracing
MeSH Terms: conditions — Elbow Injuries | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgical (Experimental): Patients undergoing surgical elbow arthrolysis. Elbow Open Arthrolyses
  Interventions: Procedure: Elbow Open Arthrolyses
- non-surgical (Experimental): Patients submitted to a non-surgical rehabilitation protocol using splints Non-surgical intervention
  Interventions: Procedure: Non-surgical intervention

INTERVENTIONS:
Procedure: Elbow Open Arthrolyses — Elbow arthrolysis by posterior access
  Other Names: surgical
  Arms: surgical
Procedure: Non-surgical intervention — Rehabilitation with splinting protocols
  Arms: non-surgical

SUMMARY:
This study compares patients with post traumatic elbow stiffness and evaluate the range of motion improvement with two types of treatment: surgical release versus non-surgical rehabilitation protocol with orthoses.

DETAILED DESCRIPTION:
The study of the treatment of post-traumatic stiffness of the elbow presents numerous challenges. Due to the great variability of the types of lesions, causes and symptomatology, there are great difficulties in the homogenization of protocols and in the comparison of results between the different treatments. Patients with different levels of severity and time of stiffness, presence of arthrosis or not, and significant symptoms such as pain.

For patients with elbow stiffness without vicious consolidation, pseudoarthrosis, intra-articular synthesis material or heterotopic ossification, and who have already failed conventional therapy, basically have two treatment options. Which will be the subject of this study: surgical release or non-surgical rehabilitation protocols with orthoses.

In meta-analysis, evaluating the elbow range of motion gain with rehabilitation protocols associated with orthoses, the mean gain varies from 20º to 40º, depending on the type of orthosis used. On the other hand a systematic review evaluated movement gain with different surgical techniques. Observed a mean gain of 51º for open releases, but with higher complication rates. However, there are no comparative studies in the literature comparing this 2 types of treatment for post traumatic elbow stiffness: surgical release and non-surgical rehabilitation protocol with orthoses in patients who have already performed conventional physiotherapy with no success.

ELIGIBILITY:
Inclusion Criteria:

* Previous history of trauma that evolved with joint stiffness at the elbow
* Range of movement of the elbow less than 100º or extension deficit greater than 30º or flexion less than 130º
* More than six months from the initial trauma;
* Skeletal maturity;
* Have had previous physical therapy without the use of orthotics or continuous passive motion for at least 4 months;
* Absence of the following findings:
* Joint block, with range of motion equal to 0º;
* Neurological limb injury;
* Mental illness or inability to understand preoperative questionnaires;
* Active infection;
* Anterior infection at the elbow;
* Systemic autoimmune diseases. (Eg, systemic lupus erythematosus, rheumatoid arthritis, joint psoriasis, etc.).
* Absence of the following radiographic changes:
* Intra-articular synthesis material;
* Presence of vicious consolidation of the distal articular surface of the humerus and proximal ulna;
* Heterotopic ossification;
* Pseudoarthrosis of previous elbow fracture;
* Elbow incongruity;
* Grade III and IV arthrosis

Exclusion Criteria:

* Non-collaboration with rehabilitation program and postoperative follow-up;
* Need to use external fixator after surgical release due to joint instability;
* Death from non-intervention causes or loss of follow-up before the first functional evaluation (3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03-03 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Elbow range of motion improvement in degrees | 6 months
  The gain will be measured with a goniometer centered on the axis of rotation of the elbow by a external examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Rames M Junior, Professor, Study Chair — University of Sao Paulo
Locations (1):
- Instituto de Ortopedia e Traumatologia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No